CLINICAL TRIAL: NCT01542580
Title: A Prospective, Clinical Investigation of the Vanguard 360 Revision Knee
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: GBMET.CR.G1
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Post Traumatic Deformity; Complications; Arthroplasty; Deformity of Limb
Keywords: Revision surgery
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Vanguard SSK 360 with PS Bearing: Patients enrolled using a Vanguard SSK 360 Posterior-Stabilized (non-constrained) tibial bearing.
  Interventions: Device: Vanguard SSK 360 with PS Bearing
- Vanguard SSK 360 with PSC Bearing: Patients enrolled using a Vanguard SSK 360 Posterior-Stabilized Constrained tibial bearing.
  Interventions: Device: Vanguard SSK 360 with PSC bearing
- Vanguard DA 360: Patients enrolled using a Vanguard DA 360 component.
  Interventions: Device: Vanguard DA 360
- Vanguard 360 TiNbN Femur with PS Bearing: The Vanguard 360 TiNbN is the same system and functions in the same manner as the non-coated device.
  Interventions: Device: Vanguard 360 TiNbN Femur with PS bearing
- Vanguard 360 TiNbN Femur with PSC Bearing: The Vanguard 360 TiNbN is the same system and functions in the same manner as the non-coated device.
  Interventions: Device: Vanguard 360 TiNbN Femur with PSC bearing

INTERVENTIONS:
Device: Vanguard SSK 360 with PS Bearing — non-constrained tibial bearing
  Groups: Vanguard SSK 360 with PS Bearing
Device: Vanguard SSK 360 with PSC bearing — constrained tibial bearing
  Groups: Vanguard SSK 360 with PSC Bearing
Device: Vanguard DA 360 — Dual-articulation device, only cleared in EU
  Groups: Vanguard DA 360
Device: Vanguard 360 TiNbN Femur with PS bearing — non-constrained tibial bearing, titanium niobium nitride coated Vanguard 360 femur
  Groups: Vanguard 360 TiNbN Femur with PS Bearing
Device: Vanguard 360 TiNbN Femur with PSC bearing — constrained tibial bearing, titanium niobium nitride coated Vanguard 360 femur
  Groups: Vanguard 360 TiNbN Femur with PSC Bearing

SUMMARY:
The purpose of this study is to evaluate performance of the Vanguard 360 revision knee system utilizing offset on either the tibial component, femoral component, or both in terms of the restoration of mechanical alignment, clinical outcomes and survivorship.

DETAILED DESCRIPTION:
This investigation is being conducted on a new complete revision knee system, Vanguard 360, which incorporates:

* Fixed Bearing Knee - Vanguard SSK360 with PS Bearing and PSC Bearing
* Fixed Bearing Knee - Vanguard SSK360 TiNbN Femur with PS Bearing and PSC Bearing
* Mobile Bearing Knee - Vanguard DA360 (only being collected in Europe)

The purpose of this study is to evaluate performance of the Vanguard 360 revision knee system utilizing offset on either the tibial component, femoral component, or both in terms of the restoration of mechanical alignment, clinical outcomes and survivorship.

The efficacy and performance of the devices will be assessed by improvement of pain, function, range of motion and patient satisfaction measured pre-operatively and post-operatively. Secondary performance and safety will be determined by radiographic investigation, incidence of complications and revision rates.

Surgical techniques and patient care are to be standard for the surgeon participating in the protocol. There will be no experimental or investigational devices used. There will be no experimental or investigational surgical techniques used. The devices and products will be used in accordance with their instructions for use and/or approved labeling.

ELIGIBILITY:
Inclusion Criteria:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus or post-traumatic deformity
* Correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure
* Ability and willingness of the patient to attend follow-up visit.
* Willing to give written informed consent
* Patients are at least 18 years of age, no upper age limit, must have reached full skeletal maturity.

Exclusion Criteria:

* infection
* sepsis
* osteomyelitis

Relative Contraindications:

* An uncooperative patient or a patient with neurologic disorders who is incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair brain function
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee

Additional research-related exclusion criteria: patients who have a history of or current infection in the affected knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed the Vanguard 360 Revision Knee System
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
AMERICAN KNEE SOCIETY KNEE SCORE | 24 months postoperative
  Improvement of American Knee Society Knee Score between pre-operative and 2 years post-operative follow up

SECONDARY OUTCOMES:
Survivorship | 10 years postoperative
  Survivorship at 10 years post-operative follow up

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (12):
- United States (4):
  - Illinois Bone and Joint, Morton Grove, Illinois
  - Orthopedic Institute of Henderson, Henderson, Nevada
  - University of Utah Orthopedic Center, Salt Lake City, Utah
  - OrthoVirginia West End Orthopedic Clinic, Richmond, Virginia
- University Hopital Pellenberg, Pellenberg, Belgium
- Aarhus university hospital, Aarhus, Denmark
- Ch Lyon Sud, Lyon, France
- Klinik fur Endoprothetik und gelenkchirurgie, Bad Wildbad, Germany
- Italy (2):
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- University Hospital Mutua de Terrasa, Terrassa, Spain
- Royal Orthopaedic Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No